CLINICAL TRIAL: NCT06996912
Title: A Phase 2 Study Investigating the Efficacy and Safety of HSK44459 Tablet Administered to Participants With Atopic Dermatitis
Brief Title: A Study for HSK44459 in Participants With Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xizang Haisco Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK44459-203
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK44459-Dose level 1 (Experimental): Participants will receive HSK44459 for 12 weeks
  Interventions: Drug: HSK44459
- HSK44459-Dose level 2 (Experimental): Participants will receive HSK44459 for 12 weeks
  Interventions: Drug: HSK44459
- Placebo (Placebo Comparator): Participants will receive Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK44459 — HSK44459 will be administered orally twice daily
  Arms: HSK44459-Dose level 1; HSK44459-Dose level 2
Drug: Placebo — Placebo will be administered orally twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of HSK44459 in adults with Atopic Dermatitis

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel group, placebo controlled phase 2 study to assess the efficacy and safety of HSK44459 in adult participants with Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Male or female, ≥18 years old and ≤75 years old
* Willing and able to comply with study-specific procedures and the requirements of this study protocol.
* Atopic dermatitis has been present for at least 1 year and subject meets Hanifin and Rajka criteria
* EASI score≥16 at the screening and baseline visits
* IGA score≥3 at the screening and baseline visits
* ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits
* Baseline WI-NRS≥4
* History of inadequate response to TCS of medium to higher potency (with or without topical calcineurin inhibitors [TCI]) or systemic treatment for AD within 6 months prior to screening
* Have applied a stable dose of topical emollient (moisturizer) twice daily for at least 7 days before the baseline visit

Exclusion Criteria:

* Subjects have used AD treatments within the time frame specified in protocol prior to the baseline visit
* Prior exposure to any PDE4 inhibitor systemic treatment
* Systemic use of known strong CYP3A inhibitors or strong CYP3A inducers within 4 weeks or 5 half-lives prior to randomization or during the course of the study
* Participation in other clinical studies within 4 weeks or 5 half-lives prior to randomization
* Subjects have laboratory values meeting the criteria in protocol
* Presence of skin comorbidities that may interfere with study assessments
* Concurrent conditions and history of other diseases as described in protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline to week 12 in EASI | From Day 1 (first dose) to Day 85 (week 12)
  Evaluate the clinical efficacy of 2 dose levels of HSK44459, compared to placebo, in adult participants with atopic dermatitis (AD) using EASI.
  A total EASI score range from 0 to 72 points will be recorded for each assessment, with higher scores reflecting worse severity of AD

SECONDARY OUTCOMES:
Proportion of patients with EASI-75 at week 12 | From Day 1 (first dose) to Day 85 (week 12)
  Proportion of patients with EASI-75 (≥75% improvement from baseline) at week 12
Proportion of patients with both IGA 0 to 1and a reduction from baseline of ≥2 points at week 12 | From Day 1 (first dose) to Day 85 (week 12)
  The IGA determines severity of AD and clinical response to treatment on a 5-point scale
  0 = Clear
  1. = Almost clear
  2. = Mild
  3. = Moderate
  4. = Severe
Proportion of patients with reduction of pruritus WI-NRS ≥3 or WI-NRS ≥4 from baseline to week 12 | From Day 1 (first dose) to Day 85 (week 12)
  The WI-NRS ranges from 0 = "no itch" to 10 ="worst imaginable itch" for the worst intensity itch in the preceding 24-hour period.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Dermatology Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No